CLINICAL TRIAL: NCT01302379
Title: Obesity-related Mechanisms and Mortality in Breast Cancer Survivors
Brief Title: Reach for Health Study: Obesity-related Mechanisms and Mortality in Breast Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Ruth E. Patterson, Professor, Department of Family & Preventive Medicine, University of California, San Diego
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Prevention
Other Study IDs: U54 CA155435-01 Project 3; U54CA155435-01 (NIH)
Record Dates: First submitted 2011-02-23; First posted 2011-02-24 (Estimated); Results first posted 2020-06-05 (Actual); Last update posted 2020-06-05 (Actual); Status verified 2020-05

CONDITIONS: Breast Neoplasms
Keywords: Obesity; Survival; Weight loss; Metformin; Biological markers
MeSH Terms: conditions — Breast Neoplasms; Obesity; Weight Loss | interventions — Metformin; Sugars

STUDY DESIGN:
Intervention Model Description: Main effects of the factorial design were the planned primary analysis and what the study was powered on.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Metformin + lifestyle intervention (Active Comparator)
  Interventions: Drug: Metformin; Behavioral: Lifestyle intervention
- Placebo + lifestyle intervention (Active Comparator)
  Interventions: Drug: Placebo; Behavioral: Lifestyle intervention
- Metformin + standard dietary guidelines (Active Comparator)
  Interventions: Drug: Metformin; Behavioral: Standard printed dietary guidelines
- Placebo + standard dietary guidelines (Placebo Comparator)
  Interventions: Drug: Placebo; Behavioral: Standard printed dietary guidelines

INTERVENTIONS:
Drug: Metformin — Week 1: 500 mg at dinner time Weeks 2-4: 1000 mg at dinner time Weeks 5+: 500 mg in morning; 1000 mg at dinner time
  Arms: Metformin + lifestyle intervention; Metformin + standard dietary guidelines
Drug: Placebo — Week 1: 1 pill at dinner time Weeks 2-4: 2 pills at dinner time Weeks 5+: 1 pill in morning; 2 pills at dinner time
  Other Names: Sugar pill
  Arms: Placebo + lifestyle intervention; Placebo + standard dietary guidelines
Behavioral: Lifestyle intervention — Telephone-based lifestyle intervention (dietary change and physical activity) for weight loss.
  Arms: Metformin + lifestyle intervention; Placebo + lifestyle intervention
Behavioral: Standard printed dietary guidelines — Set of standard health education materials provided to participants at single time point (immediately after randomization)
  Arms: Metformin + standard dietary guidelines; Placebo + standard dietary guidelines

SUMMARY:
This objective of this randomized controlled trial is to conduct a 2x2 test of a lifestyle intervention and metformin (a drug used to treat diabetes) to investigate how these treatments, alone or in combination, affect biomarkers associated with breast cancer survival. The Reach for Health Study will enroll 340 overweight/obese, postmenopausal breast cancer survivors. After completing the screening process and baseline measures, participants will be randomized in equal numbers to: (1) placebo, (2) metformin, (3) lifestyle intervention and placebo, or (4) lifestyle intervention and metformin. The intervention was powered on the main effects and the planned analyses are to compare: Metformin to Placebo and a separate comparison of Lifestyle intervention to control. The interventions will last for 6 months. Concentrations of circulating biomarkers will be assessed at baseline and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* BMI at least 25.0 kg/m2
* Diagnosed with Stage I, II, or III breast cancer within past 5 years
* Treatment with total mastectomy or breast-sparing surgical removal of cancer with clear macroscopic margins, and axillary dissection, followed by adjuvant breast radiation
* Not scheduled for or currently undergoing chemotherapy
* Accessible geographically and by telephone
* Able to communicate dietary and physical activity data via telephone
* If taking statins, tamoxifen, or aromatase inhibitors; able and willing to remain on treatment for 6-month study period
* Post-menopausal at diagnosis

Exclusion Criteria:

* Preliminary bloodwork outside of specified ranges
* Evidence of renal insufficiency, liver disease, or congestive heart failure
* Currently taking corticosteroid pills or steroid hormone therapy (including vaginal estrogen creams)
* Recent initiation (< 3 months ago) of thiazides or β-blockers
* Taking insulin or other antidiabetic drug
* Other primary or recurrent invasive cancer in past 10 years
* Unable to commit to study requirements

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 333 (Actual)
Dates: Start 2011-08; Primary Completion 2015-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Moores UCSD Cancer Center, La Jolla, California, United States

REFERENCES:
- [Derived] Bellerba F, Chatziioannou AC, Jasbi P, Robinot N, Keski-Rahkonen P, Trolat A, Vozar B, Hartman SJ, Scalbert A, Bonanni B, Johansson H, Sears DD, Gandini S. Metabolomic profiles of metformin in breast cancer survivors: a pooled analysis of plasmas from two randomized placebo-controlled trials. J Transl Med. 2022 Dec 29;20(1):629. doi: 10.1186/s12967-022-03809-6. PMID 36581893
- [Derived] Nwanaji-Enwerem JC, Chung FF, Van der Laan L, Novoloaca A, Cuenin C, Johansson H, Bonanni B, Hubbard AE, Smith MT, Hartman SJ, Cardenas A, Sears DD, Herceg Z. An epigenetic aging analysis of randomized metformin and weight loss interventions in overweight postmenopausal breast cancer survivors. Clin Epigenetics. 2021 Dec 17;13(1):224. doi: 10.1186/s13148-021-01218-y. PMID 34920739

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Metformin + Lifestyle Intervention | Placebo + Lifestyle Intervention | Metformin + Standard Dietary Guidelines | Placebo + Standard Dietary Guidelines
Started | 83 | 83 | 84 | 83
Completed | 76 | 78 | 80 | 79
Not Completed | 7 | 5 | 4 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Metformin + Lifestyle Intervention | Placebo + Lifestyle Intervention | Metformin + Standard Dietary Guidelines | Placebo + Standard Dietary Guidelines | Total
Number analyzed (Participants) | 83 | 83 | 84 | 83 | 333
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.1 (7.1) | 62.9 (62.1) | 62.1 (6.3) | 63.1 (7.4) | 62.6 (6.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 83 | 83 | 84 | 83 | 333
  Male | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 12 | 4 | 12 | 38
  Not Hispanic or Latino | 72 | 71 | 80 | 71 | 294
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 69 | 68 | 70 | 70 | 277
  Black or African American | 3 | 2 | 5 | 2 | 12
  Asian | 3 | 0 | 1 | 2 | 6
  Mixed Race or Other race | 8 | 13 | 8 | 9 | 38
Time Since Diagnosis [Mean (Standard Deviation); unit: years] | 2.4 (1.9) | 3.1 (2.4) | 2.6 (1.9) | 2.5 (1.7) | 2.7 (2.0)
Body Mass Index [Mean (Standard Deviation); unit: kg/m2] | 31.4 (5.2) | 30.8 (4.6) | 30.8 (4.7) | 31.5 (5.4) | 31.1 (5.0)

OUTCOME MEASURES:

1. Primary Outcome: Insulin
Description: Insulin measured as percent change from baseline
Time Frame: change from baseline to 6 months
Population: Obese or overweight postmenopausal breast cancer survivors
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change from baseline
Arm/Group | Metformin + Lifestyle Intervention | Placebo + Lifestyle Intervention | Metformin + Standard Dietary Guidelines | Placebo + Standard Dietary Guidelines
Number analyzed (Participants) | 83 | 83 | 84 | 83
percent change from baseline | -21.8 [-29.7 to -13.0] | -17.7 [-25.9 to -8.6] | -13.2 [-21.7 to -3.7] | -1.1 [-10.9 to 9.8]

2. Primary Outcome: Glucose
Description: Glucose measured as percent change from baseline
Time Frame: change from baseline to 6 months
Population: Obese or overweight postmenopausal breast cancer survivors
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change from baseline
Arm/Group | Metformin + Lifestyle Intervention | Placebo + Lifestyle Intervention | Metformin + Standard Dietary Guidelines | Placebo + Standard Dietary Guidelines
Number analyzed (Participants) | 83 | 83 | 84 | 83
percent change from baseline | -1.2 [-3.9 to 1.5] | -2.3 [-4.9 to 0.4] | -1.6 [-4.2 to 1.0] | 2.0 [-0.7 to 4.8]

3. Primary Outcome: C-reactive Protein
Description: C-reactive protein measured as percent change from baseline
Time Frame: change from baseline to 6 months
Population: Obese or overweight postmenopausal breast cancer survivors
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change from baseline
Arm/Group | Metformin + Lifestyle Intervention | Placebo + Lifestyle Intervention | Metformin + Standard Dietary Guidelines | Placebo + Standard Dietary Guidelines
Number analyzed (Participants) | 83 | 83 | 84 | 83
percent change from baseline | -21.4 [-38.9 to 1.0] | -6.7 [-27.4 to 19.7] | -9.2 [-29.0 to 16.1] | 5.9 [-17.4 to 35.7]

4. Primary Outcome: Bioavailable Testosterone
Description: Bioavailable testosterone measured as percent change from baseline
Time Frame: change from baseline to 6 months
Population: Obese or overweight postmenopausal breast cancer survivors
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change from baseline
Arm/Group | Metformin + Lifestyle Intervention | Placebo + Lifestyle Intervention | Metformin + Standard Dietary Guidelines | Placebo + Standard Dietary Guidelines
Number analyzed (Participants) | 83 | 83 | 84 | 83
percent change from baseline | -13.7 [-20.3 to -6.5] | -4.5 [-11.7 to 3.4] | -11.1 [-17.8 to -3.9] | -1.3 [-8.7 to 6.7]

5. Primary Outcome: Serum Hormone Binding Globulin
Description: Serum hormone binding globulin measured as percent change from baseline
Time Frame: change from baseline to 6 months
Population: Obese or overweight postmenopausal breast cancer survivors
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change from baseline
Arm/Group | Metformin + Lifestyle Intervention | Placebo + Lifestyle Intervention | Metformin + Standard Dietary Guidelines | Placebo + Standard Dietary Guidelines
Number analyzed (Participants) | 83 | 83 | 84 | 83
percent change from baseline | 12.5 [5.9 to 19.6] | 7.6 [1.4 to 14.3] | 9.8 [3.5 to 16.5] | -0.1 [-5.9 to 6.1]
Statistical Analysis 1: Comparison: Metformin + Lifestyle Intervention vs Placebo + Lifestyle Intervention vs Metformin + Standard Dietary Guidelines vs Placebo + Standard Dietary Guidelines; Test type: Superiority; p < 0.05, Mixed Models Analysis — No adjustment for multiple comparisons; Mean Difference (Final Values) = 1, 95% CI 2-sided [-97.5 to 97.5]

ADVERSE EVENTS:
Time Frame: Across the 6 month intervention
Description: The study was designed and powered for a main effects analysis and therefore the results are presented as per the original statistical plan: Metformin vs. Placebo and Lifestyle intervention vs. Control.
Groups:
- Metformin vs Placebo: Main effect for Metformin vs Placebo
- Lifestyle vs. Control: Main effect for the lifestyle intervention vs control intervention
Arm/Group | Metformin vs Placebo | Lifestyle vs. Control
Serious Adverse Events (participants affected / at risk) | 5/333 | 5/333
Other Adverse Events (participants affected / at risk) | 1/333 | 1/333
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Metformin vs Placebo (N=333) | Lifestyle vs. Control (N=333)
Injury due to fall (General disorders) | 1 (1) | 1 (1)
Abdominal pain (General disorders) | 1 (1) | 1 (1)
slurred speach (General disorders) | 1 (1) | 1 (1)
transient neurological defect (General disorders) | 1 (1) | 1 (1)
transient ischemic attack (Cardiac disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Metformin vs Placebo (N=333) | Lifestyle vs. Control (N=333)
Itching (General disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No